CLINICAL TRIAL: NCT01141374
Title: Analysis of the Application of Different Forms in Auriculotherapy on Nursing Professional Stress Levels
Brief Title: Application of Auriculotherapy on Nursing Professional Stress Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonice Fumiko Sato Kurebayashi, Leonice Fumiko Sato Kurebayashi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SISNEP
Record Dates: First submitted 2010-06-04; First posted 2010-06-10 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Stress
Keywords: Stress
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group without treatment (No Intervention): Control Group didn't receive any treatment and was evaluated at the same time and the same way of interventions group
- Auriculotherapy by needles (Experimental): The investigators used 3 points, Shenmen, Kidney, and Brain Stem with semi-permanent needles of 1.8 mm, 1 time per week for 8 sessions.
  Interventions: Other: auriculotherapy by needles
- Auriculotherapy by seeds (Experimental): The investigators used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.
  Interventions: Other: auriculotherapy by seeds

INTERVENTIONS:
Other: auriculotherapy by needles — The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.
  Other Names: auricular acupuncture
  Arms: Auriculotherapy by needles
Other: auriculotherapy by seeds — We used the three points Shenmen, Kidney, and Brain Stem with mustard seeds, 1 time per week for 8 sessions.The subjects were instructed to stimulate the points three times a day.
  Other Names: Auricular acupuncture by seeds
  Arms: Auriculotherapy by seeds

SUMMARY:
Objectives: Randomized controlled trial aimed to assess stress levels in nursing staff and review the auriculotherapy effectiveness through semi-permanent needles and seeds.

DETAILED DESCRIPTION:
Seventy five participants with average and high scores on the Stress Symptoms List (LSS) were divided in 3 groups (control, needles and seeds).

They were evaluated at the baseline, fourth and eighth sessions and 15-day follow-up and received 8 sessions through Shenmen, Kidney and Brainstem points.

ELIGIBILITY:
Inclusion Criteria:

* Average and high score by the List of Stress Symptoms
* Voluntary participation in the study
* Availability of time for submission to the sessions

Exclusion Criteria:

* Pregnancy
* Medical license or vacation during the period
* Low score of stress

Ages: 23 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Julia P Silva, Study Director — Escola de Enfermagem da Universidade de São Paulo
Locations (1):
- Hospital Universitário da Universidade de São Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted between January and July 2010 at University Hospital. Study participants were professionals from different sectors of the hospital after the invitation and 109 people answered the first questionnaire of stress (LSS). Obeying the exclusion criteria, 75 subjects were enrolled and randomized into three groups.
Pre-assignment Details: Withdrawal:employees went on vacation(7),sick leave(2), lost treatment for loss of time, forgetfulness,difficulty of rescheduling (12), withdrawal due to side effects, in this case, nightmares (1); low score (1), not belonging to the nursing staff (3), failure to attend the first session (7) not having completed the questionnaires (1)
Groups:
- Auriculotherapy by Seeds: Auriculotherapy Group by seeds at Shenmen,kidney and brainstem points,all of them for stress reduction. These points were used 1 time per week for 8 weeks. The subjects were instructed to carry out stimulation 3 times a day for at least 15 times.
- Auriculotherapy by Needles: Auriculotherapy with semi-permanent needles of 1.8mm, at shenmen, kidney and brainstem points 1 time per week for 8 weeks.
- Control Group: untreated group
Period: Overall Study
Arm/Group | Auriculotherapy by Seeds | Auriculotherapy by Needles | Control Group
Started | 26 | 27 | 22
Completed | 26 | 27 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy by Seeds | Auriculotherapy by Needles | Control Group | Total
Number analyzed (Participants) | 26 | 27 | 22 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 22 | 75
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.57 (6.40) | 41.37 (8.23) | 39.25 (13.17) | 42.06 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 21 | 71
  Male | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Brazil | 26 | 27 | 22 | 75
score stress [Mean (Standard Deviation); unit: scores on a scale] — The List of Symptoms of Stress is an evaluation questionnaire which consists of a list of 60 psycho-physiological and psychosocial stress, in which the subject must associate to each symptom of the four answers: never (0), rarely (1 ), often (2) or always (3). The scores are added together and the answers provide the level of stress the individual.In this questionnaire to score from 0 to 11 is void, 12 to 29 (low level), 30 to 59 (medium level), 60 to 120 (high level) and above 120, very high level. Participants below 29 points were excluded.
  scores on a scale | 63.27 (26.05) | 66.82 (18.56) | 54.36 (15.90) | 61.48 (20.17)

OUTCOME MEASURES:

1. Primary Outcome: Stress Levels After 4 Sessions (2nd Evaluation)
Description: Scale information: Stress Symptoms List (LSS)with 60 items (better outcome)Low score: 12/29 points; Medium score: 30/60 points; High score: 61/120 points; Very high score (worse outcome): >120 points.
Time Frame: after 30 days
Population: Of the 109 subjects, four were eliminated for having a low level of stress and 3 for not belonging to nursing staff. Of the 105, 7 didn't appear in the first session. Some lost sessions and were also excluded. One abandoned the treatment because of the side effects, one did not complete the questionnaire, seven went on vacation or sick leave (2).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: Without intervention
- Needle Group: Subjects received needles at shenmen, kidney and brainstem points, 1 time per week, during 4 weeks (2nd evaluation).
- Seeds Group: They received auriculotherapy by seeds at shenmen, kidney and brainstem points, 1 time per week, during 4 weeks (2nd evaluation).
Arm/Group | Control Group | Needle Group | Seeds Group
Number analyzed (Participants) | 22 | 27 | 26
units on a scale | 49.68 (17.99) | 54.69 (27.10) | 54.00 (25.04)
Statistical Analysis 1: Comparison: Control Group vs Needle Group vs Seeds Group; Null hypothesis: there was no statistical difference among 3 groups (control, needles and seeds) after 4 auriculotherapy sessions; Test type: Superiority or Other; p = 0.352, ANOVA — The test of hypothesis was conducted with repeated measures ANOVA with Post hoc. It was performed parametric test to compare data and the statistical significance was p<0.05; Mean Difference (Final Values) = -8.0667, 95% CI 2-sided [-76.00 to 23.00], Standard Deviation 17.28

2. Secondary Outcome: Stress Levels(3rd and 4th Evaluation)
Description: Scale Information: Stress Symptoms List (LSS) with 60 items Low score (better outcome): 12/29 points; Medium score: 30/60 points; High score: 61/120 points; Very high score (worse outcome): >120 points.
Time Frame: after 60 and 75 days
Population: 75 participants were assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Needle Group: Subjects received needles at shenmen, kidney and brainstem points, 1 time per week, during 8 weeks (3rd evaluation) and follow-up (4th evaluation).
- Seeds Group: They received auriculotherapy by seeds at shenmen, kidney and brainstem points, 1 time per week, during 8 weeks (3rd evaluation) and follow-up (4th evaluation).
Arm/Group | Control Group | Needle Group | Seeds Group
Number analyzed (Participants) | 22 | 27 | 26
units on a scale
  3rd evaluation | 67.87 (25.73) | 59.84 (23.04) | 67.10 (23.77)
  follow-up | 72.62 (31.51) | 55.54 (25.26) | 69.20 (30.03)
Statistical Analysis 1: Comparison: Control Group vs Needle Group vs Seeds Group; It was carried out the analysis of variance (ANOVA) among the groups in the 3rd assessment (after 60 days and 8 sessions). The main objective was to compare the difference among the control group, seeds and needles and to recognize significant outcomes of auriculotherapy by seeds or needles; Test type: Superiority or Other; p = 0.023, ANOVA — It was verified the normality of data distribution and the homogeneity of variance; As for the comparison between the scores, we used ANOVA for repeated measures.It was made post hoc to find the differences among groups; Mean Difference (Final Values) = -7.9067, 95% CI 2-sided [-67.00 to 37.00], Standard Deviation 19.21

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Auriculotherapy by Seeds | Auriculotherapy by Needles | Control Group
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/22
Other Adverse Events (participants affected / at risk) | 1/26 | 3/27 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auriculotherapy by Seeds (N=26) | Auriculotherapy by Needles (N=27) | Control Group (N=22)
abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — nightmares
allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — itching and redness in the auricular points
increase apettite (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — anxiety for food
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — complaints of anxiety and unrest

LIMITATIONS AND CAVEATS:
Study limitations: small sample size

Bias procedure with auricular seeds: the non-participation of the subject of research in self-massage of the points

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The copyright of the search results are the exclusive property of the Journal of School Nursing, University of Saint Paul, barring any reproduction, in whole or in part in any form or means of printed or electronic, without the prior and necessary authorization is requested.